CLINICAL TRIAL: NCT04151238
Title: Exercise Intervention for Cancer Patients to Increase Physical Activity During Chemotherapy
Brief Title: Exercise Intervention for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Turku AMK Master School (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: T306/2019
Record Dates: First submitted 2019-10-14; First posted 2019-11-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental): The duration of the exercise intervention is eight (8) weeks. There will be guided endurance and muscle power training two (2) time weekly. The participants will also be provided with one training program per week for use at home. Data on training at home and other items of physical activity is recorded in a diary.
  Interventions: Behavioral: Exercise intervention for cancer patients to increase physical activity during chemotherapy

INTERVENTIONS:
Behavioral: Exercise intervention for cancer patients to increase physical activity during chemotherapy — The duration of the exercise intervention is eight (8) weeks. There will be guided endurance and muscle power training two (2) time weekly. The participants will also be provided with one training program per week for use at home.

SUMMARY:
Exhausting chemotherapy, adverse effects of chemotherapy and a lack of information on the benefits of physical exercise are the among the reasons for reduced physical exercise among cancer patients during chemotherapy courses. According to best current knowledge only about 10% of cancer patients in Finland are physically active during cancer treatment. In addition, only 20-30% are physically active after recovery from the treatments (Pylkkänen, 2015). There is only little awareness about the benefits of physical activity during cancer treatments. The purpose of the exercise intervention study is to increase the physical activity of patients who are on chemotherapy.

The study is a pilot trial and has no control group. Internationally, exercise interventions have been studied among cancer patients on treatment for decades. The American College of Sports Medicine (ACSM) recommends that cancer patients should have 150 minutes of endurance exercise per week and at least two bouts of muscle strength exercise per week. Consequently, the exercise intervention study will have a combination of muscle power and endurance training. To reach the weekly recommended level of exercise, the cancer patients in the study will additionally have a weekly home training program containing preferentially endurance training. A literature search shows that no studies on exercise interventions during cancer treatment have been published in Finland. Thus, this thesis carries the wider implication of increasing the general knowledge on the importance of physical activity of cancer patients.

DETAILED DESCRIPTION:
The duration of the exercise intervention is eight (8) weeks. There will be guided endurance and muscle power training two (2) time weekly. The participants will also be provided with one training program per week for use at home. Data on training at home and other items of physical activity is recorded in a diary. Before the intervention is started, an oncologist will examine the participants condition before brisk physical activity is started. Safety is an important consideration and a nurse will examine the patients before each bout of exercise. A nurse will be present during the entire time of the exercise. A physician is always available for consultations by phone.

Before the intervention starts, baseline measurements will be made in the laboratories of physical exercise in the Tyks Hospital and the Turku University of Applied Sciences. At baseline, endurance, muscle power, balance and body composition will be evaluated and recorded. Endurance will be measured with a submaximal treadmill test. Muscle power will be assessed by a dynamic elevation test, hand pressure test, the lower extremities by repeated squatting-standing and by rising to stand on the toes. Balance is measured in the specific sway platform (one leg and both legs standing). The patients will be asked to fill questionnaires on quality of life (QLQ-c30) and fatigue (FACIT-F) before and after the intervention. The patients will fill in their exercise diaries from the very moment their participation has been decided until the end of the intervention. After exercise intervention the patients also fill the feedback-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients in the age of 18-70
* in the early phase of chemotherapy
* first line chemotherapy
* active way of treating cancer
* solid tumor (breast cancer, prostata cancer, colon cancer and melanoma)
* Finnish-speaking
* z=0-1 (no aids)
* capable travelling to University hospital for 8 weeks twice a week
* normal or poor physical activity background

Exclusion Criteria:

* exercise contraindications, like severe respiratory or circulatory system disease (eg. heart attack <3)
* brain or bone metastasis
* heterogenous group (max 4 patients per cancer diagnose)
* thrombocytopenia
* leukocytopenia
* immuno-oncological treatments
* really "athlete patients"

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
physical activity changes in diary | 0 and 8 weeks,
  Does this exercise intervention model works for cancer patients to increase the amount of physical activity and to achieve the cancer patients exercise recommendations? (especially home-exercising)
questionnaire-feedback from cancer patients | 0 and 8 weeks
  Does this exercise intervention model works for cancer patients to change the amount of physical activity? Patients subjective feedback about the first exercise group model in special health care. The questions are formed in quantitative way.

SECONDARY OUTCOMES:
Quality of life questionnaire (EORTC QLQ-c30) | 0 and 8 weeks
  Does the guided exercise intervention (physical activity) affect the patients quality of life during chemotherapy? The scales and single-item measures range in score from 0 to 100. High score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems. The scale consists of three different part.
Fatigue questionnaire (FACIT-F) | 0 and 8 weeks
  Does the guided exercise intervention (physical activity) affect the patients fatigue during chemotherapy? The score range: 0-52 points. The bigger points the worse fatigue or more symptoms.
Body composition in cancer patients general view (In-Body-device) | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in the body composition of cancer patients on chemotherapy? The device measures body mass index, fluid, fat and muscle changes. We follow up the changes in general view.
Endurance (submaximal treadmill test) | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in endurance of cancer patients on chemotherapy?
Functional muscle power test - dynamic elevation test for upper arms | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in muscle power of cancer patients on chemotherapy?
Functional muscle power test - hand pressure test | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in muscle power of cancer patients on chemotherapy?
Functional muscle power test - the lower extremities by repeated squatting-standing | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in muscle power of cancer patients on chemotherapy?
Functional muscle power test - the lower extremities by rising to stand on the toes | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in muscle power of cancer patients on chemotherapy?
Functional muscle power test - plank-test for the body | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in muscle power of cancer patients on chemotherapy?
Balance -tests in specific sway-platform (standing with both legs and only one leg in sway-platform) | 0 and 8 weeks
  Does exercise intervention (physical activity) cause changes in the balance of cancer patients on chemotherapy?

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No